CLINICAL TRIAL: NCT06416501
Title: The Impact of Colorectal Cancer Screening on Surgical Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, professor, Fudan University
Other Study IDs: FudanUcf
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prognosis; Colorectal Cancer; Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- screening: Patients who were detected through any screening test were categorized into the screening group
  Interventions: Other: Mode of detection
- nonscreening: Patients who were detected based on symptoms formed the non-screening group.

INTERVENTIONS:
Other: Mode of detection — Mode of detection
  Groups: screening

SUMMARY:
This study aims to investigate the pathological characteristics and surgical outcomes of stage III CRC patients detected through screening.

Data extracted from the database included the following patient information: age at diagnosis, gender, tumor location, neoadjuvant therapy, surgical procedures, histologic type, differentiation, vascular invasion, perineural invasion, pathological T stage, pathological N stage, and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent radical surgery for CRC, had confirmed stage III CRC through postoperative pathology, had no prior history of cancer before surgery, and had clear cancer detection information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent surgical intervention for CRC at Fudan University Shanghai Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-05-11 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
overall survival | the duration from the initial treatment to either death from any cause or the last recorded follow-up, whichever came first. Assessed up to 100 months.
  The duration from the initial treatment to either death from any cause or the last recorded follow-up, whichever came first.
  Assessed up to 100 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinxiang Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes